CLINICAL TRIAL: NCT02053649
Title: Integrated Chronotherapy for Perinatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: The Depressive and Bipolar Disorder Alternative Treatment Foundation (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Katherine M. Sharkey, Associate Professor, Principal Investigator, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 540053-2; 1R34MH104377-01A1 (NIH)
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Depression; Major Depressive Disorder; Postpartum Depression
Keywords: depression; major depressive disorder; postpartum depression; antenatal depression; sleep; circadian; bright light
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Usual Care will consist of medication administered by a perinatal psychiatrist and/or psychotherapy
  Interventions: Other: Usual Care
- Triple Chronotherapy + Usual Care (Experimental): triple chronotherapy (TC) will consist of bright light therapy, sleep phase advance, and sleep deprivation/restriction
  Interventions: Behavioral: Triple Chronotherapy; Other: Usual Care

INTERVENTIONS:
Behavioral: Triple Chronotherapy — triple chronotherapy (TC will consist of bright light therapy, sleep phase advance, and sleep deprivation/restriction
  Arms: Triple Chronotherapy + Usual Care
Other: Usual Care — UC will consist of medication administered by a perinatal psychiatrist and/or psychotherapy

SUMMARY:
Perinatal depression is a common and serious mood disorder that increases morbidity and mortality in new mothers and results in poor infant/child outcomes. Current therapies often fail to produce recovery or are poorly tolerated and many pregnant women seek non-pharmacologic therapy or forgo treatment when non-pharmacologic options are not available. Expectant and new mothers who suffer from circadian rhythm disruption are at risk for perinatal depression. This R34 Pilot Effectiveness Studies and Services Research Grant seeks to test whether an Integrated Chronotherapy (IC) intervention can be implemented in an outpatient psychiatry setting to improve treatment outcomes for patients with perinatal depression. IC is a multicomponent treatment consisting of bright light therapy, sleep phase advance, and sleep stabilization/restriction that targets the Research Domain Criteria (RDoC) constructs of circadian rhythms, sleep-wake behavior, social rhythms, and arousal. We will assess the feasibility, safety, and acceptability of an IC intervention for perinatal depressin by testing the treatment in expectant mothers diagnosed with major depressive disorder during 3rd trimester of pregnancy. We will randomize patients to either: (a) usual care (UC, n = 20) or (b) IC+UC (n = 20). IC+UC will have pregnancy and postpartum components and will be administered via an individualized case formulation approach tailored to each patient. After a baseline assessment, IC will be prescribed during 5 dedicated clinical visits: three during 3rd trimester of pregnancy and 2 in the postpartum period. UC will consist of medication administered by a perinatal psychiatrist and/or psychotherapy. UC will be quantified in both groups to evaluate differences between the IC+UC and UC groups. Mood will be measured in both groups by blinded clinician interview and patient self-report. We will assess the safety profile of the IC intervention with evaluation of side effects/adverse events. Importantly, the study will also examine the putative mechanisms by which IC is hypothesized to work and the "dose" of IC received by patients in the IC+UC group. All participants will wear wrist actigraphy/light monitors continuously during weeks 28-40 of pregnancy and postpartum weeks 2-6 to assess light exposure and sleep duration and timing. Circadian phase (measured with salivary dim light melatonin onset) will be measured at baseline during pregnancy (~30 weeks gestation), at 36 weeks gestation, and at postpartum week 6. This pilot will allow us to refine the IC intervention for future integration into various clinical settings and establish an infrastructue for a larger (R01-scale) trial, including measuring acceptability of IC among UC clinicians and implementing web-based data collection to facilitate data sharing in the planned R01. Perinatal IC could have major public health impact due to the high prevalence of perinatal depression and its negative effects on mothers and their children. This project represents a first step toward achieving this goal, as it will provide the pilot data necessary to prepare for a larger scale intervention study focused on providing non-pharmacologic therapies and improving outcomes for women with perinatal depression.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with a diagnosis of major depressive disorder at 24-28 weeks gestation

Exclusion Criteria:

* active psychosis or suicidality contraindicating outpatient treatment
* bipolar disorder
* seizure disorder
* self report of frequent migraines/headaches precipitated by bright light or sleep deprivation
* preexisting eye/skin disorders contraindicating light therapy
* use of photosensitizing medications
* primary Axis I diagnosis other than MDD (comorbid phobia, generalized or social anxiety disorder allowed)
* high risk pregnancy (e.g., conditions requiring mandatory bed rest or complex medical regimens that will interfere with study participation or conditions where poor infant outcomes are anticipated)
* starting antidepressants within 4 weeks of enrollment
* current employment as shift worker
* current alcohol or drug use disorders
* women whose infants will not be living in the home or who will have a nighttime caregiver
* Pittsburgh Sleep Quality Inventory (PSQI) < 5 (i.e., those who report no sleep complaints during 3rd trimester of pregnancy and for whom an intervention targeting sleep might not be indicated).
* women who do not speak and read English (because the complexity of translating the research instruments is beyond the scope of this project)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Depression Score | Change in depression score from 28 weeks of pregnancy to 6 weeks postpartum
  17-item Hamilton Depression score

SECONDARY OUTCOMES:
Sleep/Circadian Behavior | Change in Sleep/Circadian Rhythms from 28 weeks pregnancy to 6 weeks postpartum
  sleep will be measured with wrist actigraphy and circadian phase will be measured with melatonin onset

OTHER OUTCOMES:
Side Effects | Pregnancy weeks 33, 36; postpartum weeks 2, 6, 26
  Systematic Assessment for Treatment Emergent Effects

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Sharkey, MD, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Miriam Hospital Women's Medicine Collaborative, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided